CLINICAL TRIAL: NCT06994000
Title: Caring Under Pressure: The Relationship of Caregivers' Stress, Mental Health, and Self-Efficacy in ADHD Households
Brief Title: Caregiver Stress, Mental Health, and Self-Efficacy in ADHD Households
Acronym: Stress
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Assistant Professor, Alexandria University
Other Study IDs: 607/46/4838
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-02

CONDITIONS: ADHD
Keywords: Stress; Mental Health; Self-Efficacy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Descriptive Group: A convenience sample of 160 participants included caregivers of children diagnosed with ADHD (inattention, hyperactivity, or a combination thereof) by a psychiatrist, following the DSM-5 TR diagnostic criteria at neurodevelopmental centers in Saudi Arabia

SUMMARY:
Investigate the relationship between caregiver stress, mental health, and self-efficacy in families with children who have ADHD.

DETAILED DESCRIPTION:
A cross-sectional design was utilized, involving 160 caregivers from the Abdullah Al-Tamimi Autism Center in Unaizah, Saudi Arabia. Participants completed an online questionnaire that assessed sociodemographic information, caregiver stress (via the Kingston Caregiver Stress Scale), mental health (using the Mental Health Continuum-Short Form), and self-efficacy (measured by the General Self-Efficacy Scale).

ELIGIBILITY:
Inclusion Criteria:

mothers, fathers, or grandparents who are involved in the child's primary care and are between the ages of 18 and 60

Exclusion Criteria:

Caregivers who declined to participate in the current study, those who failed to complete the questionnaire, individuals not residing in the same household, and those not engaged in direct patient care

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A convenience sample of 160 participants included caregivers of children diagnosed with ADHD
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Caregiver Stress | 3 months
  This study evaluates the perceived stress levels of family caregivers during the caregiving process, as developed by Kilik and Hopkins(13). This ten-item scale has been categorized into three distinct domains: caregiving (items one to seven), family issues (items eight and nine), and financial problems (item ten). The caregiving domain gauges stress from a lack of confidence in caregiving abilities, expected future care needs of the relative, and feeling overwhelmed.
Mental Health Continuum | 3 months
  Utilizing the Multi-Item Checklist for Mental Health (MHC-SF), devised by Keyes et al. (2005)(15), this study meticulously investigated the emotional, social, and psychological (3,5,6 items, respectively) dimensions of the participants' health, serving as a self-reporting instrument for mental health assessment.
General Self-Efficacy | 3 months
  The first edition, which had 20 items, was developed in 1997; it was then reduced to 10. Since its initial development in German, the GSE scale has undergone translations into additional languages(19). The GSES was adapted to assess individuals' perceptions of personal competence. The ten items in the updated version are graded on a 4-point scale, with one denoting "not true about me" and four denoting "totally true about me."

CONTACTS AND LOCATIONS:
Locations (1):
- Qassim University, Al Qassim, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No